CLINICAL TRIAL: NCT03168230
Title: Impact of Portal Vein Embolization on Patient's Long-term Survival, Complications and Cancer Recurrence.
Brief Title: Impact of PVE on Patient's Long-term Survival, Complications and Cancer Recurrence.
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 12.106
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Liver Cancer; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVE: Patients who required PVE prior to the attempt of liver resection.
  Interventions: Procedure: Portal vein embolization (PVE)
- No-PVE: Patients who received upfront surgery (no PVE prior to the intervention)

INTERVENTIONS:
Procedure: Portal vein embolization (PVE) — Portal vein embolization (PVE) is a procedure that induces regrowth on one side of the liver in advance of a planned hepatic resection on the other side. The procedure is frequently used in primary liver cancer (hepatocellular carcinoma) and colorectal liver metastases.
  An interventional radiologist will place a needle percutaneously (through the skin) into the liver and identify the blood vessel on the side where the largest part of the tumor is being supplied. Tiny microspheres are then infused into the portal vein which supplies blood to the area, embolizing it by cutting off its blood supply.
  This blockade of the blood supply induces the other side of the liver to regrow. After several weeks, the non-embolized side has grown enough so that surgery is now a viable option.
  Source of this information : http://general.surgery.ucsf.edu/conditions--procedures/portal-vein-embolization-(pve).aspx
  Groups: PVE

SUMMARY:
For patients with colorectal liver metastasis (CLM), the prospect of long-term survival relies on liver resection. Wistfully, more than 75 % of patients with CLM are initially unresectable, due to an insufficient future liver remnant (FLR) volume

In order to increase FLR volume, most patients will first receive chemotherapy to reduce the tumor load (downsizing).

When chemotherapy is insufficient to provide an adequate postoperative FLR, portal vein embolization (PVE) can be performed. About 50-70 % of patients undergoing PVE obtain a sufficient liver hypertrophy to allow liver resection.

While PVE is recognised for its efficacy to induce liver hypertrophy, some studies expressed substantial concerns regarding the potential adverse effect of this intervention on pre-resection tumor progression, increased risk of cancer recurrence following resection and reduced overall survival following resection

Those studies suggested that the need to perform PVE should be assessed thoroughly for each patient and that chemotherapy should be maintained during the whole hypertrophy process in order to contain the potential adverse effect of PVE on tumor progression.

Other studies found no significant association between PVE and negative oncological outcomes.

As mentioned in almost every study cited above, more data is needed to provide a clearer vision regarding the impact of PVE on tumor progression and cancer recurrence following liver resection.

The aim of this study is to compare the overall and disease-free survival of PVE-requiring patients to the ones who underwent upfront surgery (NoPVE).

As a secondary objective, the impact of several covariates (related to surgery, patient's condition and disease stage) on survival and cancer recurrence will be tested.

Our hypothesis are that 1) PVE might be associated with a lower overall survival and a higher risk of cancer recurrence in univariate analysis but 2) this association will not remain significant when other covariates are included in the proportional COX hazard models.

ELIGIBILITY:
Patients with the following inclusion criterias were approached:

* Diagnosis of colorectal liver metastasis (CLM).
* Scheduled for a one-stage right/extended right hepatectomy in Centre Hospitalier Universitaire de Montréal (CHUS) - Hospital Saint-Luc.

Exclusion Criterias:

* Individuals requiring a two-stage hepatectomy.
* Patient who had previous hepatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) affected by colorectal liver metastasis (CLM) and scheduled for a one-stage right/extended right hepatectomy in Centre Hospitalier Universitaire de Montréal (CHUS) - Hospital Saint-Luc.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2004-02-27 (Actual); Primary Completion 2016-05-21 (Actual); Study Completion 2016-05-21 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
Disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yves Collin, MD, Principal Investigator — Université de Sherbrooke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collin Y, Pare A, Belblidia A, Letourneau R, Plasse M, Dagenais M, Turcotte S, Martel G, Roy A, Lapointe R, Vandenbroucke-Menu F. Portal vein embolization does not affect the long-term survival and risk of cancer recurrence among colorectal liver metastases patients: A prospective cohort study. Int J Surg. 2019 Jan;61:42-47. doi: 10.1016/j.ijsu.2018.11.029. Epub 2018 Dec 8. PMID 30537548